CLINICAL TRIAL: NCT00804713
Title: Screening for Latent Tuberculosis Infection (LTBI) in US Army Recruits
Acronym: LTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: IDCRP-021
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Latent Tuberculosis Infection
Keywords: TB; tuberculosis diagnosis; TB screening
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All study participants received 4 tests, including the use of two skin tests, one on each arm. However, the participant and outcomes assessors were blinded to which skin test was placed on which arm to avoid bias in assessment of the outcomes.
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Subjects administered the TB skin test, Battey skin test, QFT-GIT, and T-Spot
  Interventions: Drug: BST; Drug: TST; Other: QFT; Other: T-spot

INTERVENTIONS:
Drug: BST — 0.1 mcg/mL (1 dose) Battey skin test (BST) antigen administered using the Mantoux method.
Drug: TST — Administer TB Skin test (TST)
Other: QFT — Perform QFT TB test
  Other Names: Quantiferon Gold-in-tube (QFT)
Other: T-spot — Perform T-Spot TB test
  Other Names: T-spot.TB test

SUMMARY:
The overall objective of this study is to assess the feasibility and potential impact of using a targeted testing approach and 2 interferon-gamma release assays (IGRA) to screen for latent tuberculosis (TB) infection (LTBI) among military recruits. The current policy of universal application of the Mantoux tuberculin skin test (TST) to screen for LTBI may result in many TST reactions among recruits who are at low risk for LTBI. The central hypothesis is that targeted testing by use of the questionnaire will reduce unnecessary testing of low-risk recruits without affecting the identification of higher-risk recruits. The secondary hypothesis is that many discordant results between the TST and IGRA may be explained by cross-reactivity to non-tuberculous mycobacteria (NTM) with the TST.

ELIGIBILITY:
Inclusion Criteria:

* Any recruit, age 18 years or older, undergoing routine entry-level medical processing at Fort Jackson

Exclusion Criteria:

* If they have history of severe reactions to TST (e.g., blistering, scar, or symptoms of immediate hypersensitivity)
* If they are unwilling to provide written consent for the study
* If they are unwilling to provide Health Insurance Portability and Accountability Act (HIPAA) authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2017 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Mancuso, MD MPH, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Fort Jackson, SC, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Mancuso JD, Tribble D, Mazurek GH, Li Y, Olsen C, Aronson NE, Geiter L, Goodwin D, Keep LW. Impact of targeted testing for latent tuberculosis infection using commercially available diagnostics. Clin Infect Dis. 2011 Aug 1;53(3):234-44. doi: 10.1093/cid/cir321. PMID 21765072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 participants were enrolled but lost to follow-up before skin testing or blood draw were performed. This was due to the administrative requirements of the basic training setting, not because of the study itself.
Groups:
- All Study Participants: Subjects administered the tuberculosis skin test (TST), Battey skin test, Quantiferon Gold-in-tube (QFT-GIT), and T-Spot
Period: Overall Study
Arm/Group | All Study Participants
Started | 1978
Completed | 1978
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: recruits at Fort Jackson, SC in 2009 between April 1 and June 11
Groups:
- All Study Participants: Subjects administered the Tuberculosis skin test (TST), Battey skin test, QFT-GIT, and T-spot
Arm/Group | All Study Participants
Number analyzed (Participants) | 1978
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (4.6)
Sex/Gender, Customized [Number; unit: participants] — sex of participants. The number doesn not equal 1978 because of missing responses on the questionnaire.
  participants
    Female | 681
    Male | 1294
Prevalence of tuberculosis (TB) in country of birth [Number; unit: participants] — Prevalence of TB per 100,000 population
  participants
    <20 per 100,000 | 1811
    20-99 per 100,000 | 62
    >=100 per 100,000 | 105

OUTCOME MEASURES:

1. Primary Outcome: TST Induration Will be Interpreted Relative to Risk, in Accordance With Published CDC Guidelines.
Description: Risk stratification and test result. Risk was stratified by the use of risk factors identified by questionnaire according to the 5, 10 and 15 mm criteria (CDC Morbidity and Mortality Weekly Report Recommendations and Reports 2000. Targeted Testing for Latent Tuberculosis Infection.)
  The number of 1803 is used here because that is the number for which valid results were available for all 4 tests.
  The number presented in each category is the number of participants that had positive results.
  We are only presented a risk stratified interpretation for the TST (not the QFT, T-spot, and BST) because that is the only test for which this methodology is accepted in scientific and medical use. It is also the only test for which we had pre-specified the use of this methodology in the protocol.
Time Frame: 48-72 hrs post administration
Measure: Number; unit: participants
Groups:
- All Study Participants: Subjects administered the TB skin test
  Tuberculin Skin Test: Administer TB Skin test, Battey skin test, QFT, and T-Spot
Arm/Group | All Study Participants
Number analyzed (Participants) | 1803
participants
  High | 2
  Medium | 37
  Low | 20

2. Secondary Outcome: Positive QFT-GIT Result
Description: The number of subjects is 1781 (less than the original 1978) because we analyzed only those who had valid results by all 4 tests to have a fair comparison. Additionally, we excluded those subject who had a borderline T-Spot result, as we were not able to make valid comparisons with these results.
Time Frame: 48-72 hours after enrollment
Measure: Number; unit: participants
Groups:
- QFT-GIT: Subjects administered the QFT-GIT TB test
  QFT-GIT: Perform QFT-GIT TB test
Arm/Group | QFT-GIT
Number analyzed (Participants) | 1781
participants
  Positive | 36
  Negative | 1745

3. Other Pre Specified Outcome: T-Spot Result
Description: Positive T-Spot results. The number of subjects is 1781 (less than the original 1978) because we analyzed only those who had valid results by all 4 tests to have a fair comparison. Additionally, we excluded those subject who had a borderline T-Spot result, as we were not able to make valid comparisons with these results.
Time Frame: 48-72 hours
Measure: Number; unit: participants
Groups:
- All Study Participants: Subjects administered the TB skin test, Battey skin test, QFT-GIT, and T-Spot
  All study participants: 0.1 mcg/mL (1 dose) Battey skin test antigen administered using the Mantoux method.
  All study participants: Administer TB Skin test
  All study participants: Perform QFT-GIT TB test
  All study participants: Perform T-Spot TB test
Arm/Group | All Study Participants
Number analyzed (Participants) | 1781
participants
  Positive | 34
  Negative | 1747

4. Other Pre Specified Outcome: Battey Skin Test Result
Description: Battey skin test positive results defined as >= 100 mm reaction. The number of subjects is 1781 (less than the original 1978) because we analyzed only those who had valid results by all 4 tests to have a fair comparison. Additionally, we excluded those subject who had a borderline T-Spot result, as we were not able to make valid comparisons with these results.
Time Frame: 48-72 hours after administration
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 1781
participants
  Positive | 203
  Negative | 1578

5. Other Pre Specified Outcome: TST Results for the Population for Which All 4 Tests Have Valid Results and no Borderline Results
Time Frame: 48-72 hours after adminstration
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 1781
participants
  Positive | 48
  Negative | 1733

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/1978
Other Adverse Events (participants affected / at risk) | 0/1978

LIMITATIONS AND CAVEATS:
A limitation of this study is the lack of a gold standard for determining the presence of M. tuberculosis infection, making it difficult to assess the true significance of discordance between TST and the interferon-gamma release assays (IGRAs).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No